CLINICAL TRIAL: NCT03767231
Title: Emergency Department Patient's Perceptions and Acceptability Toward a Novel Point-of-Care Hepatitis C Virus Viral Load Testing
Brief Title: ED Patient's Perceptions and Acceptability Toward a Novel POC HCV Viral Load Testing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Cepheid (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00171078
Record Dates: First submitted 2018-12-05; First posted 2018-12-06 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Hepatitis C
Keywords: viral load testing; point of care
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HCV POC VL Group (Experimental): This group will receive the POC HCV viral load testing via fingerstick using the novel Xpert HCV Viral Load Finger-stick Point-of-Care test (Cepheid) in addition to the standard-of-care whole-blood conventional laboratory-based HCV PCR viral load testing. Participants in this group will also fill out a short survey regarding participant's socio-demographic information as well as participant's experience, attitudes, and perceptions regarding HCV testing and care.
  Interventions: Diagnostic Test: Xpert HCV Viral Load Finger-stick Point-of-Care test (Cepheid)
- Reference Group (No Intervention): This group will receive the standard-of-care whole-blood conventional laboratory-based HCV PCR viral load testing only. Participants in this group will also fill out a short survey regarding participant's socio-demographic information as well as participant's experience, attitudes, and perceptions regarding HCV testing and care.

INTERVENTIONS:
Diagnostic Test: Xpert HCV Viral Load Finger-stick Point-of-Care test (Cepheid) — The investigators will randomly assign eligible and consented patients to either to HCV POC VL Group or Reference Group. All participants will take a short survey regarding HCV care and treatment. As part of the investigators' ED HCV Screening and Linkage to Care Program, all participants will receive the standard-of-care clinical laboratory-based HCV RNA viral load testing via whole blood (i.e. patient will receive blood drawn). This standard-of-care HCV viral load testing result will be provided to participant when it is available (usually 1-2 days later). Participants in the HCV POC VL Group will receive the novel POC HCV RNA viral load testing and the result of the novel test will be disclosed to the patients approximately within 1 to 1½ hours of the testing.
  Arms: HCV POC VL Group

SUMMARY:
Hepatitis C virus (HCV) infection has become the leading fatal infectious disease in the United States. Approximately 75% of individuals who have been infected with HCV are chronically infected with the virus. Untreated chronic infection will lead to severe sequelae such as cirrhosis and hepatocellular carcinoma. Even though the availability of rapid HCV antibody (HCV Ab) screening assay and highly effective antiviral treatment, most people infected with HCV are not aware of the infection status. This gap mainly comes from the current gold standard confirmatory testing for chronic HCV infection, the Polymerase Chain Reaction (PCR)-based HCV RNA viral load assay which requires an experienced trained laboratory technician to perform relatively complicated PCR assay with a turn-around-time of 1 to 2 days (from provider's order to the test resulting). The investigators' rapid HCV Screening and Linkage to Care program has demonstrated that many patients in the investigators' emergency department (ED) are unaware of patient's chronic HCV infection status due to the barriers to receive the gold standard viral load testing.

Recently, a novel Xpert HCV Viral Load (VL) Finger-stick (FS) [Xpert HCV VL FS] point-of-care (POC) test (Cepheid) has been developed. In an observational cohort in Australia, HCV RNA was detected in 40% of participants (85 of 210) enrolled at 3 drug treatment clinics and 1 homelessness service. Sensitivity of the Xpert HCV VL FS assay for HCV RNA quantification in samples collected by finger-stick was 100.0% (95% Confidence Interval (CI), 93.9%-100.0%) and specificity was 100.0% (95% CI, 96.6%-100.0%). The Xpert HCV VL FS test can accurately detect active infection from a finger-stick sample in 1 hour allowing single-visit HCV diagnosis.

In this protocol, the investigators seek to determine the needs and acceptability of a novel POC HCV viral load testing assay among ED HCV Ab positive patients. For this project, the investigators will identify and enroll ED patients with HCV Ab positive but without HCV viral information. The investigators will conduct a randomized study to assign eligible and consented patients to either to POC Testing Group or Standard of Care (SOC) Group. All participants will take a short survey regarding HCV care and treatment. As part of the investigators' ED HCV Screening and Linkage to Care Program, all participants will receive the standard-of-care clinical laboratory-based HCV RNA viral load testing via whole blood (i.e. patient will receive blood drawn). This standard-of-care HCV viral load testing result will be provided to participant when it is available (usually 1-2 days later). Participants in the POC Testing Group will receive the novel POC HCV RNA viral load testing and the result of the novel test will be disclosed to the patients approximately within 2 hours of the testing. Linkage to care information after the ED visit will be compared between two groups. Finally, accuracy of this POC HCV RNA viral load testing in the acute care setting will be determined as compared to the standard-of-care clinical laboratory-based HCV RNA viral load testing. The investigators will also ask all of participants to grant permission to use the remnant blood specimens for an evaluation of future in-house HCV RNA viral load assay.

DETAILED DESCRIPTION:
Johns Hopkins Emergency Department-Based Rapid HCV Screening and Linkage to Care Program

Johns Hopkins Hospital Emergency Department (JHHED) has implemented an ED-based rapid HCV Screening and Linkage to Care Program since late 2015, after adapting the 2012 Centers for Disease Control and Prevention (CDC) revised HCV testing recommendations. The investigators' program utilizes an integrated, triage nurse driven model to deliver opt-out HCV testing to eligible ED patients. Eligibility was facilitated by electronic health record (EHR) prompts to identify patients over the age of 17 years and no HCV testing history at the institution. For patients who were medically/surgically stable and who did not have altered mental status, an opt-out HCV Ab test offering was delivered by staff. JHHED utilizes the blood-based anti-HCV assay (Abbott Architect) and fingerstick POC HCV assay (OraSure) for HCV Ab testing, depending on the availability of patient's whole blood drawn for his/her ED care. HCV reflex RNA testing is performed for HCV Ab reactive patients tested by blood-based HCV Ab assay. Blood specimens for HCV RNA testing are collected during the ED visit (if possible) for HCV Ab reactive patients tested by POC HCV Ab assay with confirmatory testing performed asynchronous to the ED visit. JHHED utilized dedicated linkage to care program staff that contacted ED patients with HCV Ab reactive results to deliver confirmatory results and facilitate referral to HCV care. The investigators' program staff also identify HCV Ab positive patients without HCV RNA viral load information by screening the ED tracking board (EPIC) to inform ED providers of ordering HCV RNA viral load testing which might need to have blood drawing if there is no blood work ordered in place.

Routine Care All JHHED patients are eligible for HCV screening or linkage to care service under the investigators' ED-based rapid HCV Screening and Linkage to Care Program if participants are 18 years and older, no history of HCV diagnosis or testing, and do not have altered mental status. Please see the brief description of the investigators' program above.

Recruitment A. Steps for recruiting participants with known HCV antibody positive but no HCV viral load data

1. The ED HCV Screening and Linkage to Care (LTC) Program will screen the ED tracking board (EPIC) for patients who potentially meet study enrollment criteria (i.e. not possessing any exclusion criteria), which is done routinely as a part of standard of care. The ED HCV Screening and LTC team will notify the research coordinator of all eligible patients.
2. Research coordinator will then approach the treating ED clinician for his/her patients regarding the research opportunity in the investigators' study.
3. Providers may refer eligible patients to research coordinator after getting permission from patients. Providers who are part of the investigators' study team will refer the eligible patients to research coordinator after patients agree to be approached by the investigators' research coordinator regarding the investigators' study.

For providers who are not in the investigators' study team, the recruitment procedure will be that the patient's clinician will request permission from patients and document in the chart regarding the patient's permission to be contacted by the research staff.

B. Steps for recruiting participants with newly diagnosed HCV antibody positive identified from ED HCV Screening and Linkage to Care Program

1. Research coordinator will work closely with ED HCV Screening and Linkage to Care Program staff to recruit this subgroup of ED patients. Screening Program staff will notify the research coordinator via pager (or equivalent) when an ED patient is diagnosed with HCV Ab reactive result via the Screening Program.
2. Research coordinator will then approach the treating ED clinician for his/her patients regarding the research opportunity in the investigators' study.
3. Providers may refer eligible patients to research coordinator after getting permission from patients. Providers who are part of the investigators' study team will refer the eligible patients to research coordinator after patients agree to be approached by the investigators' research coordinator regarding the study.

For providers who are not in the investigators' study team, the recruitment procedure will be that the patient's clinician will request permission from patients and document in the chart regarding the patient's permission to be contacted by the research staff.

Enrollment The research coordinator will obtain oral, informed consent. The process will involve a description of the study as provided in the verbal consent form with a chance to provide answers to any questions about the study. Justification for verbal consent is provided in the electronic Institutional Review Board (e-IRB) application. Specifically, this study poses minimal risk to patients. The consent process will take between approximately 15-20 minutes, based on the requirements of the individual patient.

Consented subjects will be given a copy of the oral consent document for participant's information and records. In this consent, the patient will be asked for permission to review patient's medical charts at Johns Hopkins Hospital for the clinical information of the ED visit and subsequent HCV-related visits. In addition, the patient will be asked for permission to allow the investigators to use the remnant blood specimen of this study in the future for an evaluation of an in-house HCV RNA viral load assay. Consented patients will be randomized to one of two groups, HCV POC Testing Group or Standard of Care (SOC) Group. The testing group will receive the POC HCV viral load testing via fingerstick using a novel Xpert HCV Viral Load Finger-stick (Xpert HCV VL FS) point-of-care (POC) test and the reference group will not receive this POC VL testing. Both groups will receive stand of care conventional laboratory-based whole blood HCV VL testing. Consented patients in both groups will fill out a short survey regarding participant's socio-demographic information as well as participant's experience, attitudes, and perceptions regarding HCV testing and care

ELIGIBILITY:
Inclusion Criteria:

* Any Johns Hopkins Emergency Department patient who has HCV antibody positive result but no HCV RNA test result in the chart
* Able to provide informed consent
* 18-100 years

Exclusion Criteria:

* Patient who has a diagnosis of chronic HCV infection
* Patient with a non-reactive test result of an HCV Ab screening test
* Patient with a chief complaint of sexual assault
* Patients who are otherwise ineligible to consent due to medical condition (e.g., severe illness, altered mental status)
* Any person who has previously enrolled in this study
* Any person less than 18 years of age
* Any person who is incarcerated
* Any woman who is pregnant
* Any person who is transgender
* Any person who is sex worker
* Any person who is refugee

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-11 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Acceptability of POC HCV viral load testing as assessed by a Likert scale | At the time of enrollment, up to 15 minutes
  The acceptability will be assessed using the 5-point Likert Scale (1-5) with scores of 3 or higher indicating acceptability. There will be one question for this outcome.
Linkage to care rates between the HCV POC VL group and the control group | 12 months
  Percentage of patients who receive standard of care HCV viral load testing entering care for HCV and percentage of patients who receive POC HCV viral load testing in the ED entering care for HCV will be calculated and used in the assessment of linkage to care rate.

SECONDARY OUTCOMES:
Accuracy of an in-house POC HCV viral load assay (developed by Dr. Tza-Huei Wang) as assessed by sensitivity of the assay | 12 months
  Sensitivity of the in-house POC HCV viral load assay will be determined by the proportion of true positives that are identified as such by the assay.
Accuracy of an in-house POC HCV viral load assay (developed by Dr. Tza-Huei Wang) as assessed by specificity of the assay | 12 months
  Specificity of the in-house POC HCV viral load assay will be determined by the proportion of true negatives that are identified as such by the assay.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Hsiang Hsieh, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith BD, Morgan RL, Beckett GA, Falck-Ytter Y, Holtzman D, Teo CG, Jewett A, Baack B, Rein DB, Patel N, Alter M, Yartel A, Ward JW; Centers for Disease Control and Prevention. Recommendations for the identification of chronic hepatitis C virus infection among persons born during 1945-1965. MMWR Recomm Rep. 2012 Aug 17;61(RR-4):1-32. PMID 22895429
- [Background] Grebely J, Applegate TL, Cunningham P, Feld JJ. Hepatitis C point-of-care diagnostics: in search of a single visit diagnosis. Expert Rev Mol Diagn. 2017 Dec;17(12):1109-1115. doi: 10.1080/14737159.2017.1400385. Epub 2017 Nov 8. PMID 29088981
- [Background] Rein DB, Wittenborn JS, Weinbaum CM, Sabin M, Smith BD, Lesesne SB. Forecasting the morbidity and mortality associated with prevalent cases of pre-cirrhotic chronic hepatitis C in the United States. Dig Liver Dis. 2011 Jan;43(1):66-72. doi: 10.1016/j.dld.2010.05.006. Epub 2010 Jun 17. PMID 20739252
- [Background] Brillman JC, Crandall CS, Florence CS, Jacobs JL. Prevalence and risk factors associated with hepatitis C in ED patients. Am J Emerg Med. 2002 Sep;20(5):476-80. doi: 10.1053/ajem.2002.32642. PMID 12216048
- [Background] Galbraith JW, Franco RA, Donnelly JP, Rodgers JB, Morgan JM, Viles AF, Overton ET, Saag MS, Wang HE. Unrecognized chronic hepatitis C virus infection among baby boomers in the emergency department. Hepatology. 2015 Mar;61(3):776-82. doi: 10.1002/hep.27410. Epub 2015 Jan 28. PMID 25179527
- [Background] Hsieh YH, Rothman RE, Laeyendecker OB, Kelen GD, Avornu A, Patel EU, Kim J, Irvin R, Thomas DL, Quinn TC. Evaluation of the Centers for Disease Control and Prevention Recommendations for Hepatitis C Virus Testing in an Urban Emergency Department. Clin Infect Dis. 2016 May 1;62(9):1059-65. doi: 10.1093/cid/ciw074. Epub 2016 Feb 21. PMID 26908800
- [Background] Kelen GD, Green GB, Purcell RH, Chan DW, Qaqish BF, Sivertson KT, Quinn TC. Hepatitis B and hepatitis C in emergency department patients. N Engl J Med. 1992 May 21;326(21):1399-404. doi: 10.1056/NEJM199205213262105. PMID 1373867
- [Background] Lyons MS, Kunnathur VA, Rouster SD, Hart KW, Sperling MI, Fichtenbaum CJ, Sherman KE. Prevalence of Diagnosed and Undiagnosed Hepatitis C in a Midwestern Urban Emergency Department. Clin Infect Dis. 2016 May 1;62(9):1066-71. doi: 10.1093/cid/ciw073. Epub 2016 Feb 21. PMID 26908799
- [Background] Anderson ES, Galbraith JW, Deering LJ, Pfeil SK, Todorovic T, Rodgers JB, Forsythe JM, Franco R, Wang H, Wang NE, White DAE. Continuum of Care for Hepatitis C Virus Among Patients Diagnosed in the Emergency Department Setting. Clin Infect Dis. 2017 Jun 1;64(11):1540-1546. doi: 10.1093/cid/cix163. PMID 28207069
- [Background] McHugh MP, Wu AHB, Chevaliez S, Pawlotsky JM, Hallin M, Templeton KE. Multicenter Evaluation of the Cepheid Xpert Hepatitis C Virus Viral Load Assay. J Clin Microbiol. 2017 May;55(5):1550-1556. doi: 10.1128/JCM.02460-16. Epub 2017 Mar 8. PMID 28275079
- [Background] Pinsky BA, Sahoo MK, Sandlund J, Kleman M, Kulkarni M, Grufman P, Nygren M, Kwiatkowski R, Baron EJ, Tenover F, Denison B, Higuchi R, Van Atta R, Beer NR, Carrillo AC, Naraghi-Arani P, Mire CE, Ranadheera C, Grolla A, Lagerqvist N, Persing DH. Analytical Performance Characteristics of the Cepheid GeneXpert Ebola Assay for the Detection of Ebola Virus. PLoS One. 2015 Nov 12;10(11):e0142216. doi: 10.1371/journal.pone.0142216. eCollection 2015. PMID 26562786
- [Background] Mahilum-Tapay L, Laitila V, Wawrzyniak JJ, Lee HH, Alexander S, Ison C, Swain A, Barber P, Ushiro-Lumb I, Goh BT. New point of care Chlamydia Rapid Test--bridging the gap between diagnosis and treatment: performance evaluation study. BMJ. 2007 Dec 8;335(7631):1190-4. doi: 10.1136/bmj.39402.463854.AE. Epub 2007 Nov 30. PMID 18055487
- [Background] Shin DJ, Trick AY, Hsieh YH, Thomas DL, Wang TH. Sample-to-Answer Droplet Magnetofluidic Platform for Point-of-Care Hepatitis C Viral Load Quantitation. Sci Rep. 2018 Jun 28;8(1):9793. doi: 10.1038/s41598-018-28124-3. PMID 29955160
- [Background] Bajis S, Maher L, Treloar C, Hajarizadeh B, Lamoury FMJ, Mowat Y, Schulz M, Marshall AD, Cunningham EB, Cock V, Ezard N, Gorton C, Hayllar J, Smith J, Whelan M, Martinello M, Applegate TL, Dore GJ, Grebely J; LiveRLife Study Group. Acceptability and preferences of point-of-care finger-stick whole-blood and venepuncture hepatitis C virus testing among people who inject drugs in Australia. Int J Drug Policy. 2018 Nov;61:23-30. doi: 10.1016/j.drugpo.2018.08.011. Epub 2018 Oct 25. PMID 30388566
- [Background] Fekete T. The Xpert HCV Viral Load Finger-Stick point-of-care test was accurate for detecting HCV RNA. Ann Intern Med. 2018 Sep 18;169(6):JC35. doi: 10.7326/ACPJC-2018-169-6-035. No abstract available. PMID 30242408
- [Background] Lamoury FMJ, Bajis S, Hajarizadeh B, Marshall AD, Martinello M, Ivanova E, Catlett B, Mowat Y, Marks P, Amin J, Smith J, Ezard N, Cock V, Hayllar J, Persing DH, Kleman M, Cunningham P, Dore GJ, Applegate TL, Grebely J; LiveRLife Study Group. Evaluation of the Xpert HCV Viral Load Finger-Stick Point-of-Care Assay. J Infect Dis. 2018 May 25;217(12):1889-1896. doi: 10.1093/infdis/jiy114. PMID 29534185
- [Background] Grebely J, Lamoury FMJ, Hajarizadeh B, Mowat Y, Marshall AD, Bajis S, Marks P, Amin J, Smith J, Edwards M, Gorton C, Ezard N, Persing D, Kleman M, Cunningham P, Catlett B, Dore GJ, Applegate TL; LiveRLife Study Group. Evaluation of the Xpert HCV Viral Load point-of-care assay from venepuncture-collected and finger-stick capillary whole-blood samples: a cohort study. Lancet Gastroenterol Hepatol. 2017 Jul;2(7):514-520. doi: 10.1016/S2468-1253(17)30075-4. Epub 2017 Apr 22. PMID 28442271
- See also: Hepatitis C - Fact Sheet. World Health Organization, 2017. — http://www.who.int/mediacentre/factsheets/fs164/en/